CLINICAL TRIAL: NCT02325505
Title: Clinical Profile Characterization of Patients With Tuberous Sclerosis Complex, Lymphangioleiomyomatosis and Angiomyolipoma Followed at Hospital Das Clínicas, University of Sao Paulo Medical School
Brief Title: Characterization of Patients With Tuberous Sclerosis Complex, Lymphangioleiomyomatosis and Angiomyolipoma
Status: Completed | Type: Observational
Sponsor: InCor Heart Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Bruno Guedes Baldi, Medical Assistant, InCor Heart Institute
Other Study IDs: 4147/14/127
Record Dates: First submitted 2014-12-14; First posted 2014-12-25 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Tuberous Sclerosis; Lymphangioleiomyomatosis; Angiomyolipoma
MeSH Terms: conditions — Tuberous Sclerosis; Lymphangioleiomyomatosis; Angiomyolipoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tuberous sclerosis complex: All patients with TSC, LAM or AML followed at Hospital das Clínicas, University of São Paulo Medical School will be included in the proposed study. Patients of all ages will participate in the study.

SUMMARY:
Tuberous Sclerosis Complex (TSC) is a multisystemic autosomal dominant disease that is characterized by the development of benign neoplasms in brain, kidney, lung, skin and heart. TSC is caused by mutations in TSC1 and/or TSC2 genes, which encode, respectively, hamartin and tuberin, that are involved in the regulation of cell proliferation, cell cycle and protein synthesis. Most patients exhibit dermatological, renal, neurological and pulmonary (lymphangioleiomyomatosis, LAM) manifestations. Neurological involvement include subependymal nodules, subependymal giant cell astrocytomas and cortical tubers. LAM is characterized by the proliferation of LAM cells around the airways, blood vessels and lymphatics, which result in vascular and airway obstruction and cyst formation. The most frequent TSC manifestation in the kidney is the development of angiomyolipomas (AML). Dermatologic lesions represent the most common manifestations of TSC, mainly hypomelanotic macules and facial angiofibromas. The most significant functional implication of the tuberin-hamartin complex is its regulatory role upon the mammalian target of rapamycin (mTOR) pathway. Mutations in TSC1 or TSC2 lead to increased mTOR activity and favor tumor development and growth. All lesions associated with TSC, sporadic LAM and sporadic AML share a common molecular pathogenesis, based on TSC1/TSC2 mutations and mTOR hyperactivity. Up to date, TSC patients have been followed in separated medical services in our institution, according to their predominant phenotype. The current knowledge, however, suggest that the ideal follow up of such patients should be conducted in an integrated fashion among the specialties associated with the main disease manifestations. Experts in TSC from each of these areas have recently created a TSC/LAM/AML integrated program in the University of São Paulo Medical Center, and his project will be initiated with the generation of an integrated TSC/LAM/AML registry, which intends not only to clinically characterize this patient population but also to document the employed treatment modalities. Once this first goal is achieved, clinical trials are planned to be performed. The central aim of this observational study is to clinically characterize the TSC/LAM/AML subject population followed and referred to the University of São Paulo Medical Center. Specific aims: To characterize the pulmonary, the neurological, the renal and the dermatologic phenotypes of this patient population.

DETAILED DESCRIPTION:
1. Introduction Tuberous Sclerosis Complex (TSC) is a multisystemic autosomal dominant disease , that is characterized by the development of histologically benign neoplasms in brain, kidney, lung, skin, heart and eyes, as well as by central nervous system (CNS) disorganization. TSC is caused by mutations in TSC1 (Tuberous Sclerosis Complex 1) and/or TSC2 genes, which encode, respectively, hamartin and tuberin, proteins that form a complex involved in the regulation of cell proliferation, cell cycle and protein synthesis. Although the majority of organs are susceptible, most patients exhibit dermatological, renal, neurological and pulmonary manifestations.

   Involvement of the CNS responds for most of TSC morbidity and include subependymal nodules, subependymal giant cell astrocytomas (SEGA) and cortical tubers, alterations prone to lead to ventricular obstruction, hydrocephalus, epilepsy, intellectual disability and psychiatric problems.

   Lymphangioleiomyomatosis (LAM) is a rare disease that is characterized by the proliferation of LAM cells around the airways, blood vessels and lymphatics, which can result in vascular and airway obstruction and cyst formation. LAM occurs sporadically or in association with tuberous sclerosis complex. The main clinical features are dyspnea, pneumothorax and chylothorax.

   The most frequent TSC manifestation in the kidney is the development of angiomyolipomas (AML), a tumor derived from perivascular epithelioid cells that comprises abnormally organized blood vessels, smooth muscle cells and adipose tissue. AML affects 60-80% of TSC patients, but it also occurs sporadically. The main AML-related complication is renal hemorrhage, the most common cause of mortality in adults with TSC.

   Dermatologic lesions represent the most common manifestations of TSC, mainly hypomelanotic macules and facial angiofibromas.

   The most significant functional implication of the tuberin-hamartin complex is its regulatory role upon the mammalian target of rapamycin (mTOR) pathway. Mutations in TSC1 or TSC2 lead to increased mTOR activity and favor tumor development and growth. Interestingly, all lesions associated with TSC, sporadic LAM and sporadic AML share a common molecular pathogenesis, based on TSC1/TSC2 mutations and mTOR hyperactivity.

   A number of studies have shown potentially beneficial effects of mTOR inhibitors on LAM and TSC patients with SEGA and AML, including sirolimus and everolimus. Such positive effects, however, are heterogeneous among these manifestations and critical pieces of information are lacking to define the true roles of mTOR inhibitors on each of TSC manifestations, as well as the sporadic forms of LAM and AML.
2. Study rational The University of São Paulo Medical School is the main and largest medical complex in Latin America. Up to date, TSC patients have been followed in separated medical services in our institution, according to their predominant phenotype. The current knowledge and therapeutic perspectives, however, suggest that from this moment on the ideal follow up of such patients should be conducted in an integrated fashion among the specialties associated with the main disease manifestations, ie, neurology, pulmonary, nephrology, urology and dermatology. Experts in TSC from each of these areas have recently come together to create a TSC/LAM/AML integrated program in the University of São Paulo Medical School, with the aim of building a Brazilian TSC Reference Center. This center is expected to provide integrated clinical follow up of TSC patients. We also expect to bring this center to a reference status for the entire country.

   This project will be initiated with the generation of an integrated TSC/LAM/AML registry, including all TSC and LAM cases and selected AML patients according to potential severity. This database is planned to be fed and accessed by all physicians included in the current proposal. Such this registry intends not only to clinically characterize this patient population but also to document the employed treatment modalities. Once this first goal is achieved, strategic and well-designed clinical studies are planned to be performed, including clinical trials with mTOR inhibitors.
3. Objectives 3.1. Primary objective The central aim of this observational study is to clinically characterize all patients with TSC, LAM and AML followed and referred to the University of São Paulo Medical School.

   3.2. Secondary objectives

   - To characterize the pulmonary phenotype of this patient sample, by integrating conventional clinical findings with radiological and pulmonary functional test features.
   * To characterize the neurological phenotype of the analyzed patient population, by composing the clinical observations with radiological findings and surgical and post-surgery follow-ups.
   * To characterize the renal phenotype of the evaluated patient population by integrating the clinical findings with radiologic alterations and surgical and post-surgery follow-ups.
   * To characterize the dermatologic phenotype of this patient population.
   * To establish data about loss of productivity and hospitalizations during the study in the analyzed patient population.
4. Study design This is an observational study that aims to describe mainly respiratory, neurological, renal and dermatological features of the all patients with TSC, LAM or AML followed at the University of São Paulo Medical Center. The study also aims to establish the impact of these diseases on loss of productivity and also to establish data about hospitalizations during the study in the patient population. This proposal intends to expand the comprehension of TSC pathogenesis and manifestations and to create a robust platform to perform interventional clinical trials.

The flow of the current study comprises the following steps:

1. Creation of an integrated database 2. Patient selection according to the inclusion criteria 3. Data collection 4. Data analysis and assessment 5. Interpretation of results and generation of reports

5. Population The population of this study is composed of patients with TSC, LAM or AML. The estimated sample size for this study is 200 patients.

5.1. Inclusion criteria

• All patients with TSC, LAM or AML followed at Hospital das Clínicas, University of São Paulo Medical School will be included in the proposed study. Patients of all ages will participate in the study.

5.2. Exclusion criteria • There is no exclusion criteria. 6. Assessments

This study includes the following evaluations:

A) Clinical evaluation

- Demographic and anthropometric data

- Criteria for tuberous sclerosis complex (if present)

- Family history for the diseases evaluated in the study

- Previous and current treatments

- Data about loss of productivity and hospitalizations during the study

* Quality of life evaluation with the questionnaire Short-Form Health Survey - 36
* Characterization of skin lesions
* Urinary and abdominal complaints
* Previous or current smoking
* Respiratory symptoms
* Assessment of the degree of dyspnea using baseline dyspnea index B) Skin biopsy (if necessary) C) Abdominal ultrasonography D) Abdominal computed tomography or nuclear magnetic resonance (if there is a suspected or a definitive lesion identified in abdominal ultrasonography) E) Chest high resolution computed tomography F) Computed tomography or nuclear magnetic resonance of the brain G) Electroencephalogram H) Spirometry I) Pulmonary volumes and diffusion capacity for carbon monoxide (if there is any change in spirometry and/or in chest high resolution computed tomography) J) Transthoracic echocardiography K) Six-minute walking test (if there is any change in spirometry and/or in chest high resolution computed tomography) 7. Data collection and management Data will be collected and stored in a database developed specifically for this study.

  8. Statistical methods and data analysis 8.1. Sample size The estimated sample size for this study is 200 patients. All patients followed in the Neurology, Respiratory, Nephrology, Urology and Dermatology services at University of Sao Paulo Medical School will be included in the study.

9.2. Population for analysis We will analyze data about all patients included in the database. 9.3. Statistical methods Data will be presented as mean and standard deviation (or standard error) for parametric variables, defined by the normal curve on the histogram, and as median and interquartile range (IQ) for nonparametric variables. Categorical variables will be expressed as percentages.

9. Ethical aspects 9.1. Ethics and Good Pharmacoepidemiology Practices By signing the protocol, the investigator agrees to comply with the instructions described and the Good Pharmacoepidemiology Practices (GPP), the Declaration of Helsinki and other applicable regulatory requirements. The study will also be performed so that local legal requirements are met.

9.2. Institutional Review Board / Independent Ethics Committee IN PROGRESS 9.3. Informed Consent Form Eligible patients may only be enrolled in the study after providing the written informed consent (witnessed, whenever required by law or regulation), approved by the EC or, if unable to do it, after this consent is provided by an accepted legal representative of the patient. In cases in which the patient's representative provides the consent, the patient must be informed about the study as far as possible, considering his/her understanding. If the patient is able to understand, he/she must indicate his/her consent by personally signing and dating the written informed consent form or a separate consent form. Informed consent form must be obtained before the conduction of any procedure specific to the study (i.e., all the procedures described in the protocol).

9.4. Declaration of Helsinki The participant investigator should conduct the study according to the principles of the Declaration of Helsinki. Copies of the Declaration of Helsinki and amendments will be provided upon request or may be accessed through the website of the World Medical Association at http://www.wma.net/e/policy/17-c_e.html.

10. Recording of data and retention of documents Study duration: 24 months Study start : March 2015 Recruitment end: March 2016 Study end: March 2017 Follow-up: From March 2016 to March 2017 11. Study sponsorship and funding This study was fully prepared by the investigator-sponsor. The investigator-sponsor and local institution are responsible for the costs arising from this study. Novartis Biociências S.A. does not have any participation in preparation, logistics, data collection and storage, statistical evaluation, result interpretation and manuscript wording for publication. There is no type of restriction or external control by Novartis Biociências S.A. The contribution of Novartis Biociências S.A. is only intended to make viable part of the Study aspects that, otherwise, would not be feasible. The Investigator-Sponsor and the investigator institution will be in charge of insurance matters.

ELIGIBILITY:
Inclusion Criteria:

* All patients with TSC, LAM (sporadic or associated with TSC) or AML (sporadic or associated with TSC or with LAM) followed at Hospital das Clínicas, University of São Paulo Medical School will be included in the proposed study. Patients of all ages will participate in the study.

Exclusion Criteria:

* There is no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this study is composed of patients with TSC, LAM (sporadic or associated with TSC) or AML (sporadic or associated with TSC or with LAM). The estimated sample size for this study is about 200 patients, all of them followed at University of Sao Paulo Medical School.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04; Primary Completion 2021-04 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Pulmonary function tests | Baseline and change after one year
  Decline of forced expiratory volume in the first second
Chest high resolution computed tomography findings | Baseline and change after one year
  Extent of pulmonary cysts
Findings on computed tomography of the brain | Baseline and change after one year
  TSC lesions
Abdominal computed tomography findings | Baseline and change after one year
  Renal angiomyolipoma, lymphangioleiomyoma
Skin lesions | Baseline and change after one year
  Describe skin lesions in the study population
Respiratory symptoms Describe all respiratory symptoms in the study population) | Baseline and change after one year
  Describe all respiratory symptoms in the study population
Quality of life evaluation with the questionnaire Short-Form Health Survey - 36 (SF-36) | Baseline and change after one year
  Absolute variation
Urinary and abdominal complaints | Baseline and change after one year
  Describe urinary and abdominal complaints in the study population
Baseline dyspna index | Baseline and change after one year
  Assessment of the degree of dyspnea using baseline dyspnea index
Treatments performed (previous and current treatments performed) | Baseline
  To describe previous and current treatments performed
Neurological complaints | Baseline and after one year
  Describe neurological complaints in the study population

SECONDARY OUTCOMES:
Six-minute walking distance and dessaturation during six-minute walk test | Baseline and change after one year
  Variation in walking distance and oxygen saturation inone year
Systolic pulmonary arterial pressure | Baseline and after one year
  This valuable will be evaluated by transthoracic echocardiography
Histopathological characteristics of samples obtained from skin biopsy | Baseline
  If there is a skin lesion, it might be biopsied and evaluated by a pathologist

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Roberto Ribeiro Carvalho, MD, PhD, Principal Investigator — InCor Heart Institute
Locations (2):
- Brazil (2):
  - InCor Heart Institute, São Paulo
  - InCor Heart Institute, Research Center, São Paulo

REFERENCES:
- [Background] Franz DN, Bissler JJ, McCormack FX. Tuberous sclerosis complex: neurological, renal and pulmonary manifestations. Neuropediatrics. 2010 Oct;41(5):199-208. doi: 10.1055/s-0030-1269906. Epub 2011 Jan 5. PMID 21210335
- [Background] Curatolo P, Bombardieri R, Jozwiak S. Tuberous sclerosis. Lancet. 2008 Aug 23;372(9639):657-68. doi: 10.1016/S0140-6736(08)61279-9. PMID 18722871
- [Background] Crino PB, Nathanson KL, Henske EP. The tuberous sclerosis complex. N Engl J Med. 2006 Sep 28;355(13):1345-56. doi: 10.1056/NEJMra055323. No abstract available. PMID 17005952
- [Background] Franz DN, Belousova E, Sparagana S, Bebin EM, Frost M, Kuperman R, Witt O, Kohrman MH, Flamini JR, Wu JY, Curatolo P, de Vries PJ, Whittemore VH, Thiele EA, Ford JP, Shah G, Cauwel H, Lebwohl D, Sahmoud T, Jozwiak S. Efficacy and safety of everolimus for subependymal giant cell astrocytomas associated with tuberous sclerosis complex (EXIST-1): a multicentre, randomised, placebo-controlled phase 3 trial. Lancet. 2013 Jan 12;381(9861):125-32. doi: 10.1016/S0140-6736(12)61134-9. Epub 2012 Nov 14. PMID 23158522
- [Background] Datta AN, Hahn CD, Sahin M. Clinical presentation and diagnosis of tuberous sclerosis complex in infancy. J Child Neurol. 2008 Mar;23(3):268-73. doi: 10.1177/0883073807309250. Epub 2008 Jan 29. PMID 18230839
- [Background] Johnson SR, Cordier JF, Lazor R, Cottin V, Costabel U, Harari S, Reynaud-Gaubert M, Boehler A, Brauner M, Popper H, Bonetti F, Kingswood C; Review Panel of the ERS LAM Task Force. European Respiratory Society guidelines for the diagnosis and management of lymphangioleiomyomatosis. Eur Respir J. 2010 Jan;35(1):14-26. doi: 10.1183/09031936.00076209. No abstract available. PMID 20044458
- [Background] Ryu JH, Moss J, Beck GJ, Lee JC, Brown KK, Chapman JT, Finlay GA, Olson EJ, Ruoss SJ, Maurer JR, Raffin TA, Peavy HH, McCarthy K, Taveira-Dasilva A, McCormack FX, Avila NA, Decastro RM, Jacobs SS, Stylianou M, Fanburg BL; NHLBI LAM Registry Group. The NHLBI lymphangioleiomyomatosis registry: characteristics of 230 patients at enrollment. Am J Respir Crit Care Med. 2006 Jan 1;173(1):105-11. doi: 10.1164/rccm.200409-1298OC. Epub 2005 Oct 6. PMID 16210669
- [Background] Baldi BG, Albuquerque AL, Pimenta SP, Salge JM, Kairalla RA, Carvalho CR. Exercise performance and dynamic hyperinflation in lymphangioleiomyomatosis. Am J Respir Crit Care Med. 2012 Aug 15;186(4):341-8. doi: 10.1164/rccm.201203-0372OC. Epub 2012 Jun 14. PMID 22700863
- [Background] Bissler JJ, Kingswood JC, Radzikowska E, Zonnenberg BA, Frost M, Belousova E, Sauter M, Nonomura N, Brakemeier S, de Vries PJ, Whittemore VH, Chen D, Sahmoud T, Shah G, Lincy J, Lebwohl D, Budde K. Everolimus for angiomyolipoma associated with tuberous sclerosis complex or sporadic lymphangioleiomyomatosis (EXIST-2): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2013 Mar 9;381(9869):817-24. doi: 10.1016/S0140-6736(12)61767-X. PMID 23312829
- [Background] Schwartz RA, Fernandez G, Kotulska K, Jozwiak S. Tuberous sclerosis complex: advances in diagnosis, genetics, and management. J Am Acad Dermatol. 2007 Aug;57(2):189-202. doi: 10.1016/j.jaad.2007.05.004. PMID 17637444
- [Background] Roach ES, Gomez MR, Northrup H. Tuberous sclerosis complex consensus conference: revised clinical diagnostic criteria. J Child Neurol. 1998 Dec;13(12):624-8. doi: 10.1177/088307389801301206. PMID 9881533
- [Background] McCormack FX, Inoue Y, Moss J, Singer LG, Strange C, Nakata K, Barker AF, Chapman JT, Brantly ML, Stocks JM, Brown KK, Lynch JP 3rd, Goldberg HJ, Young LR, Kinder BW, Downey GP, Sullivan EJ, Colby TV, McKay RT, Cohen MM, Korbee L, Taveira-DaSilva AM, Lee HS, Krischer JP, Trapnell BC; National Institutes of Health Rare Lung Diseases Consortium; MILES Trial Group. Efficacy and safety of sirolimus in lymphangioleiomyomatosis. N Engl J Med. 2011 Apr 28;364(17):1595-606. doi: 10.1056/NEJMoa1100391. Epub 2011 Mar 16. PMID 21410393
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Mahler DA, Weinberg DH, Wells CK, Feinstein AR. The measurement of dyspnea. Contents, interobserver agreement, and physiologic correlates of two new clinical indexes. Chest. 1984 Jun;85(6):751-8. doi: 10.1378/chest.85.6.751. PMID 6723384
- [Background] Mahler DA, Harver A, Rosiello R, Daubenspeck JA. Measurement of respiratory sensation in interstitial lung disease. Evaluation of clinical dyspnea ratings and magnitude scaling. Chest. 1989 Oct;96(4):767-71. doi: 10.1378/chest.96.4.767. PMID 2791670
- [Background] Assumpcao Junior FB, Kuczynski E, Gabriel MR, Rocca CC. [Evaluation scale of autistic behavior. Validity and reliability of a scale for autistic behavior detection]. Arq Neuropsiquiatr. 1999 Mar;57(1):23-9. doi: 10.1590/s0004-282x1999000100005. Portuguese. PMID 10347719
- [Background] Santos RS, Araujo AP, Porto MA. Early diagnosis of abnormal development of preterm newborns: assessment instruments. J Pediatr (Rio J). 2008 Jul-Aug;84(4):289-99. doi: 10.2223/JPED.1815. PMID 18688553
- [Background] Miotto EC, Sato J, Lucia MC, Camargo CH, Scaff M. Development of an adapted version of the Boston Naming Test for Portuguese speakers. Braz J Psychiatry. 2010 Sep;32(3):279-82. doi: 10.1590/s1516-44462010005000006. Epub 2010 Apr 30. PMID 20428731
- [Background] Gerstadt CL, Hong YJ, Diamond A. The relationship between cognition and action: performance of children 3 1/2-7 years old on a Stroop-like day-night test. Cognition. 1994 Nov;53(2):129-53. doi: 10.1016/0010-0277(94)90068-x. PMID 7805351
- [Background] Pereira CA, Sato T, Rodrigues SC. New reference values for forced spirometry in white adults in Brazil. J Bras Pneumol. 2007 Jul-Aug;33(4):397-406. doi: 10.1590/s1806-37132007000400008. English, Portuguese. PMID 17982531
- [Background] Duarte AA, Pereira CA, Rodrigues SC. Validation of new brazilian predicted values for forced spirometry in caucasians and comparison with predicted values obtained using other reference equations. J Bras Pneumol. 2007 Sep-Oct;33(5):527-35. doi: 10.1590/s1806-37132007000500007. English, Portuguese. PMID 18026650
- [Background] Neder JA, Andreoni S, Castelo-Filho A, Nery LE. Reference values for lung function tests. I. Static volumes. Braz J Med Biol Res. 1999 Jun;32(6):703-17. doi: 10.1590/s0100-879x1999000600006. PMID 10412549
- [Background] Neder JA, Andreoni S, Peres C, Nery LE. Reference values for lung function tests. III. Carbon monoxide diffusing capacity (transfer factor). Braz J Med Biol Res. 1999 Jun;32(6):729-37. doi: 10.1590/s0100-879x1999000600008. PMID 10412551
- [Background] Soaresa MR, Pereira CA. Six-minute walk test: reference values for healthy adults in Brazil. J Bras Pneumol. 2011 Sep-Oct;37(5):576-83. doi: 10.1590/s1806-37132011000500003. English, Portuguese. PMID 22042388
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180